CLINICAL TRIAL: NCT01117701
Title: Does a Safety Guidewire Adjacent to the Ureteroscope Increase the Forces Needed to Move the Ureteroscope up and Down the Ureter?
Brief Title: Does a Safety Guidewire Increase the Forces Needed to Move the Ureteroscope up and Down the Ureter?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse-Bergen HF (Other)
Responsible Party: Øyvind Ulvik, MD, Helse Bergen HF, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 102.09 (REK) - 4; 21835 (NSD) - 4 (Other: Norway: Norwegian Social Science Data Services); 102.09 (REK) - 4 (Other: The National Committees for Research Ethics in Norway)
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2011-06

CONDITIONS: Ureteroscopy
MeSH Terms: interventions — Ureteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - with SGW (Experimental): Measurement of the forces needed to passage the ureteroscope in the ureter with a SGW in place.
  Interventions: Procedure: Ureteroscopy with and without safety guidewire
- B - without SGW (Experimental): Measurement of the forces needed to passage the ureteroscope in the ureter without a SGW in place.
  Interventions: Procedure: Ureteroscopy with and without safety guidewire

INTERVENTIONS:
Procedure: Ureteroscopy with and without safety guidewire — In study arm A - with SGW, the force measurements are made with a safety guidewire in place. In study arm B - without SGW, the force measurements are made without SGW.

SUMMARY:
The purpose of this study is to investigate to forces needed to passage the ureteroscope up and down the ureter with and without a safety guidewire in place.

DETAILED DESCRIPTION:
Ureteroscopy may damage the ureter, and the complication risk is influenced by the forces needed to move the ureteroscope up and down the ureter.

Although a safety guidewire (SGW) is commonly recommended in order to reduce the complication rate it may well be that the SGW itself may inhibit the passage of the ureteroscope due to increased friction.

The forces needed to move the ureteroscope in the ureter have not been investigated properly.

The intention in this study is to measure the forces needed to advance and withdraw the ureteroscope in the ureter with and without the SGW in place.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for endoscopic kidney stone treatment

Exclusion Criteria:

* Known pathology in the ureter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The force needed to passage the ureteroscope up and down in the ureter with and without SGW. | 1 day
  The force is measured by a digital force-meter device. The force measured is scaled in Newton. The results are available immediately after each measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Ulvik, MD, Principal Investigator — Helse Bergen HF, Haukeland University Hospital
Locations (1):
- Helse Bergen HF, Haukeland University Hospital, Bergen, Bergen, Norway